CLINICAL TRIAL: NCT01715064
Title: Acute Effects of Exercise on the Cortical Silent Period in Prostate Cancer Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Guelph-Humber (Other)
Responsible Party: Principal Investigator, Daniel Santa Mina, Assistant Program Head, Kinesiology, University of Guelph-Humber
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PCA_CSP2012
Record Dates: First submitted 2012-10-09; First posted 2012-10-26 (Estimated); Results first posted 2014-02-10 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Exercise; Cortical Inhibition; Cortical Silent Period; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): non-exercise control consisting of movie watching.
- Exercise (Experimental): 1 hour of moderate intensity exercise.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — 1 hour of moderate-intensity exercise
  Arms: Exercise

SUMMARY:
In Canadian men, prostate cancer (PCa) is the most prevalent form of cancer and the third leading cause of cancer-related death. Unfortunately, PCa survivors are often burdened with feelings of anxiety and depression associated with the disease and associated treatments. Short-term exercise interventions (8-24 weeks) have improved psychosocial well-being in this population, but the impact of single bouts of exercise and related psychological or neurological changes have never been studied. The primary objective of the proposed study is to examine the effect of an acute bout of exercise on neurophysiological and psychological indicators of well-being in a randomized controlled trial (RCT) of 36 men with PCa. Participants will be randomly assigned to the intervention (60 min exercise) or control (60 min of television) and will undergo a brief neurological test (cortical silent period) and psychological questionnaires before and after their group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed PCa;
* > 6 months post curative therapy for PCa (radical prostatectomy or radiation therapy) with or without adjuvant androgen deprivation therapy;
* Willing and able to provide informed consent;
* If metastatic disease is present, they are asymptomatic; v) n
* No contraindications to exercise

Exclusion Criteria:

* Severe coronary artery disease (Canadian Cardiovascular Society class III or greater);
* Significant congestive heart failure (New York Heart Association class III or greater);
* Uncontrolled pain;
* Neurological or musculoskeletal co-morbidity inhibiting exercise;
* Diagnosed psychotic, addictive, or major cognitive disorders or are currently or have a history of using psychotropic medication (anti-depressants, anti-anxiety, anti-psychotics, benzodiazepines, etc);
* Contraindications to magnetic exposure (surgical clips in the brain; cardiac pace maker or valves; cochlear implants; metal rods, plates, screws in head; shrapnel/metal fragments in head/eyes; dentures);
* Prior history of seizures or diagnosis of epilepsy;
* Left-hand dominant; and
* No more than two of the following Coronary Risk Factors as defined by the American College of Sports Medicine[41, 42]:

  * Family history of coronary disease, cigarette smoking, hypertension (Systolic Blood Pressure (SBP) > 140 mmHg; Diastolic Blood Pressure (DBP) > 90 mmHg), known dyslipidemia, known impaired fasting, glucose (>110 mg/dL), obesity (BMI > 30 kg/m2 or waist circumference > 102cm), or physically inactive (<150 min of moderate intensity physical activity per week)

Ages: 45 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Santa Mina D, Guglietti CL, de Jesus DR, Azargive S, Matthew AG, Alibhai SM, Trachtenberg J, Daskalakis JZ, Ritvo P. The acute effects of exercise on cortical excitation and psychosocial outcomes in men treated for prostate cancer: a randomized controlled trial. Front Aging Neurosci. 2014 Nov 26;6:332. doi: 10.3389/fnagi.2014.00332. eCollection 2014. PMID 25505413

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were approached for participation by a research coordinator from June to October, 2010. 86 eligible participants were approached for participation and 19 agreed (22% participation rate). Seventeen participants responded to the study poster. The 36 participants were randomly assigned to the exercise (n=18) or control (n=18) group.
Groups:
- Control (1hr of Viewing Emotionally Neutral Movie): non-exercise control consisting of movie watching for 60 mins. the videos were short cartoon films considered to be emotionally neutral.
- Exercise (1hr of Mixed-modality Exercise): 1 hour of moderate intensity exercise. The session included 5- min warm-up, 25-min of resistance training, 25-min of aerobic training, and 5-min cool-down. Each session was led by a personal trainer and supervised by an exercise physiologist.
Period: Overall Study
Arm/Group | Control (1hr of Viewing Emotionally Neutral Movie) | Exercise (1hr of Mixed-modality Exercise)
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Exercise | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 15 | 28
  >=65 years | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (9.1) | 67.7 (7.6) | 64.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 18 | 18 | 36
Region of Enrollment [Number; unit: participants]
  Canada | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cortical Silent Period (CSP) Will be Determined Using Transcranial Magnetic Stimulation (TMS) of the Motor Cortex.
Description: CSP is a measure of cortical inhibition that is negatively related to anxiety, stress, and depression.
Time Frame: 10-15 minutes prior to the control/exercise condition ('pre-test') and 10-15 minutes after the control/exercise condition ('post-test').
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Control | Exercise
Number analyzed (Participants) | 18 | 18
seconds | 0.001 (0.025) | 0.006 (0.019)

2. Secondary Outcome: Profile of Mood States Questionnaire(PoMS)
Description: Correlations will be assessed between cortical silent period and acute mood state.
Time Frame: as for outcome 1
Reporting Status: Not Posted

3. Secondary Outcome: State-Trait Anxiety Inventory - Questionnaire(STAI)
Description: Correlations will be assessed between cortical silent period and acute anxiety.
Time Frame: as for outcome 1
Reporting Status: Not Posted

4. Secondary Outcome: Hospital Anxiety and Depression Scale - Questionnaire(HADS)
Description: Correlations will be assessed between cortical silent period and acute anxiety and depression.
Time Frame: as for outcome 1
Reporting Status: Not Posted

5. Secondary Outcome: Exercise-Induced Feelings Inventory - Questionnaire (EIFI)
Description: Correlations will be assessed between cortical silent period and exercise-induced feelings.
Time Frame: as for outcome 1
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 7 months.
Description: Serious adverse and other adverse events were collected during participants' activity in the trial (i.e. the pre-treatment assessment, during the exercise or video sessions, and during the post-treatment assessment).
Arm/Group | Control | Exercise
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes